CLINICAL TRIAL: NCT07087756
Title: The Effect of Temporary Ovarian Suspension to the Anterior Abdominal Wall During Laparoscopic Endometriosis Surgery for Adhesion Prevention -A Comparative and Prospective Study
Brief Title: The Effect of Temporary Ovarian Suspension to the Abdominal Wall During Laparoscopic Endometriosis Surgery for Adhesion Prevention -A Comparative and Prospective Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Yuval Kaufman, Head of the Multidisciplinary Center for the Treatment of Endometriosis, Carmel Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CMC-0110-24
Record Dates: First submitted 2025-06-26; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Endometriosis; Abdominal Adhesions
Keywords: endometriosis; ovarian suspension; laparoscopy; abdominal adhesions
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suspended Ovary (Active Comparator): Ovary suspended during laparoscopy for endometriosis surgery
  Interventions: Procedure: laparoscopic ovarian suspension
- Non-suspended ovary (Sham Comparator): Ovaries not suspended during laparoscopy for endometriosis
  Interventions: Procedure: laparoscopic ovarian suspension

INTERVENTIONS:
Procedure: laparoscopic ovarian suspension — Suspension of the ovary during laparoscopy for endometriosis

SUMMARY:
Pelvic adhesions, particularly between ovaries and pelvic sidewall, frequently complicate endometriosis surgery. Despite various interventions, no widely accepted solution exists. Small studies suggest temporary ovarian suspension may reduce adhesion formation. This technique, which temporarily elevates ovaries postoperatively, shows promise but requires further investigation to confirm its efficacy and long-term outcomes.

This prospective, single-blinded, randomized controlled study compares adhesion formation in endometriosis patients at risk for ovarian adhesions. Participants are randomized to undergo laparoscopic surgery with temporary ovarian suspension or standard care without ovarian suspension. Pain and suture removal eagerness are assessed via daily questionnaires. Blinded ultrasound experts evaluate adhesions at 6 and 13 weeks postoperatively. No anti-adhesive barriers are used to minimize confounding factors

DETAILED DESCRIPTION:
Endometriosis is a chronic condition characterized by growth of endometrial tissue in sites other than the uterine cavity, most commonly in the pelvic cavity, including the ovaries, the uterosacral ligaments, and the pouch of Douglas. Laparoscopic excision of endometriosis lesions has become the gold standard treatment. At follow-up, relief of pain and quality of life after endometriosis surgical treatment ranges between 50% and 95%. However, pelvic surgery for endometriosis has been associated with a high rate of postoperative adhesion formation. The incidence of pelvic adhesions at second-look laparoscopy in the initial few weeks after surgery has been reported to be between 50% and 100%. The ovaries are the most common site involved by adhesions because of their anatomic localization (close to the pelvic sidewall and the homolateral tube) and the fragility of the coelomic epithelium that covers the ovarian surface [7,8]. In addition, when the posterior pelvic compartment is involved, obliteration of the pouch of Douglas is often observed as a result of a post-inflammatory process causing ovarian adhesions [9]. Women with higher risk for postoperative ovarian adhesions include those who have preoperative ovarian adhesions or patients undergoing ovarian cystectomy, peritonectomy of the ovarian fossa or extensive pelvic adhesiolysis. Postoperative retained free fluid with blood and postoperative infections may also increase the risk for adhesions. Postoperative adhesions are a source of major concern because of their potential consequences including persistent pelvic pain, dyspareunia (difficult or painful sexual intercourse), infertility, intestinal obstruction, and complications at subsequent surgery.

A wide range of interventions has been tried in the past in order to reduce postoperative pelvic adhesions. This includes intra-peritoneal administration of anti-adhesive solutions such as icodextrin and hyaluronic acid. Various drugs including steroids and heparin have also been tried in the past but none of them have gained wide acceptance (Metwally et al., 2006; Kamel, 2010). Oxidized regenerated cellulose was found to reduce postoperative adhesion in two very small RCTs (Ahmad et al., 2008).

Intra-operative suspension of the ovaries to the anterior abdominal wall is sometimes used to facilitate ovarian retraction and improve exposure of the pelvis during surgery for severe endometriosis (Cutner et al., 2004). Temporary ovarian suspension can be achieved using a straight needle and absorbable suture to suspend the ovary to the abdominal wall with an external knot tie that can be easily removed at any time after surgery. Two small observational studies suggested that temporary ovarian suspension for 4-7 days following surgery for severe endometriosis may reduce the frequency of postoperative pelvic adhesions (Abuzeid et al., 2002; Ouahba et al., 2004).

The Objective of the Study The primary objective of the study is to examine adhesion formation following laparoscopic surgery with temporary ovarian suspension removed a week after surgery.

The secondary objective is the analyze patient symptoms and adherence to the ovarian suspension as well as request to remove the suture before one week post operative.

Rationale for conducting the study If ovarian suspension is indeed beneficial it can be incorporated as part of common practice for laparoscopic endometriosis surgery.

Methods This is a prospective single-blinded randomized controlled interventional study.

Patients scheduled for laparoscopic surgery due to endometriosis with suspected adnexal adhesions, lesions of the ovary, ovarian fossa, uterosacral ligaments, pouch of Douglas, or involvement of the bowel, as seen by imaging, will be included. A comparison will be made between suspended ovaries in the study group vs. non-suspended ovaries in the control group. During surgery, the primary surgeon will inspect the pelvis. If on the side of the relevant ovary there are adhesions and/or ovarian cyst and/or peritoneal lesions around the ovarian fossa and uterosacral ligament, an ovarian suspension will be performed according to randomization. The randomization process will be based on a preformed list produced by the statistician which will be used during surgery. In case of bilateral pelvic involvement, the left ovary will be the first to be acted on according to the randomization result (i.e suspend/not suspend). In case of ovarian cysts, the surgeon will decide upon treatment method of the cyst during surgery. Suspension of the ovary will be performed using Monocryl absorbable suture. In order to reduce confounding variables, there will be no use of anti-adhesive barriers. Removal of the suspension will be performed at the clinic a week after surgery unless the patient requests to remove the suture earlier. Patients will be asked to fill a daily questionnaire describing the amount of pain according to VAS score they are experiencing due to ovarian suspension and how eager they are to remove the suture prematurely on a scale of 1-10.

Preoperative and postoperative ultrasound evaluation will be performed by one of two dedicated ultrasound experts using a Voluson E10 ultrasound. During postoperative evaluation, the experts will be blinded as to whether ovarian suspension was performed or not. Postoperative ultrasound will be performed 6 and 13 weeks following surgery and will include description of the size of the ovary, location and severity of adhesions.

Statistical analysis will be performed according to each suspended vs non-suspended ovary, i.e. the number of ovaries suspended for the study group vs, the number of non-suspended ovaries in the control group patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate to severe endometriosis with suspected adhesions, lesions in the ovary, ovarian fossa, utero-sacral ligaments, pouch of douglas, or involvement of the intestine as seen in preoperative assessment who are willing to participate in the study including postoperative follow-up assessments.

Exclusion Criteria:

* Patients who are not intended to have an endometriosis operation. Patients with minimal to mild endometriosis and no suspected adhesions or ovarian, ovarian fossa, utero-sacral ligament, pouch of douglas involvement on preoperative assessment.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-03-16 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Adhesion formation following laparoscopic surgery with temporary ovarian suspension as assessed in post-operative ultrasound visits at weeks 6,13 following surgery | From enrollment to last follow-up visit at 13 weeks post surgery
  The primary objective of the study is to examine adhesion formation following laparoscopic surgery with temporary ovarian suspension removed a week after surgery. Assessment of adhesions will be performed by ultrasound before surgery and then at 6 week and 13-week post-surgery. Assessment will be performed by an ultrasound specialist who is blinded to the surgical procedure. Adhesions are marked as negative or positive per organ including left and right ovary, left and right tube and other locations (rectosigmoid, uterus, bladder, pouch of Douglas).

SECONDARY OUTCOMES:
Patient pain during the first week following laparoscopy | From enrollment to 1 week post-operative follow-up visit
  The secondary objective is to analyze patient pain symptoms during the first week after surgery. Patients will report pain symptoms daily, as measured by Visual Analog Score for pain on a scale of 0-10.
Patient tolerability to ovarian suspension during the first week following surgery | From enrollment to 1 week post-operative follow-up visit
  Patient will report daily on their eagerness to remove the suture temporarily suspending each ovary to the abdominal wall on a scale from 0 to 10 during the first week after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Carmel Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Yes
Patients outcomes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data available from 26/6/2025 till study termination estimated at around 1/7/2025

REFERENCES:
- [Background] Davey AK, Maher PJ. Surgical adhesions: a timely update, a great challenge for the future. J Minim Invasive Gynecol. 2007 Jan-Feb;14(1):15-22. doi: 10.1016/j.jmig.2006.07.013. PMID 17218224
- [Background] Hudelist G, Fritzer N, Staettner S, Tammaa A, Tinelli A, Sparic R, Keckstein J. Uterine sliding sign: a simple sonographic predictor for presence of deep infiltrating endometriosis of the rectum. Ultrasound Obstet Gynecol. 2013 Jun;41(6):692-5. doi: 10.1002/uog.12431. PMID 23400893
- [Background] diZerega GS, Campeau JD. Peritoneal repair and post-surgical adhesion formation. Hum Reprod Update. 2001 Nov-Dec;7(6):547-55. doi: 10.1093/humupd/7.6.547. PMID 11727863
- [Background] Kavic SM, Kavic SM. Adhesions and adhesiolysis: the role of laparoscopy. JSLS. 2002 Apr-Jun;6(2):99-109. PMID 12113430
- [Background] diZerega GS. Contemporary adhesion prevention. Fertil Steril. 1994 Feb;61(2):219-35. doi: 10.1016/s0015-0282(16)56507-8. PMID 8299773
- [Background] Mabrouk M, Montanari G, Guerrini M, Villa G, Solfrini S, Vicenzi C, Mignemi G, Zannoni L, Frasca C, Di Donato N, Facchini C, Del Forno S, Geraci E, Ferrini G, Raimondo D, Alvisi S, Seracchioli R. Does laparoscopic management of deep infiltrating endometriosis improve quality of life? A prospective study. Health Qual Life Outcomes. 2011 Nov 6;9:98. doi: 10.1186/1477-7525-9-98. PMID 22054310
- [Background] Ouahba J, Madelenat P, Poncelet C. Transient abdominal ovariopexy for adhesion prevention in patients who underwent surgery for severe pelvic endometriosis. Fertil Steril. 2004 Nov;82(5):1407-11. doi: 10.1016/j.fertnstert.2004.03.060. PMID 15533368
- [Background] Garry R, Clayton R, Hawe J. The effect of endometriosis and its radical laparoscopic excision on quality of life indicators. BJOG. 2000 Jan;107(1):44-54. doi: 10.1111/j.1471-0528.2000.tb11578.x. PMID 10645861
- [Background] Garry R. Laparoscopic excision of endometriosis: the treatment of choice? Br J Obstet Gynaecol. 1997 May;104(5):513-5. doi: 10.1111/j.1471-0528.1997.tb11523.x. No abstract available. PMID 9166188
- [Background] Farquhar C. Endometriosis. BMJ. 2007 Feb 3;334(7587):249-53. doi: 10.1136/bmj.39073.736829.BE. No abstract available. PMID 17272567